CLINICAL TRIAL: NCT04406259
Title: Atrioventricular Block and Cluster Headache
Brief Title: Atrioventricular Block and Cluster Headache (SEVA)
Acronym: SEVA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-API-03
Record Dates: First submitted 2020-05-14; First posted 2020-05-28 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — Verapamil

STUDY DESIGN:
Intervention Model Description: prospective cohort, interventional , multicentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Verapamil (Other): administration of verapamil to treat cluster headache
  Interventions: Drug: Verapamil

INTERVENTIONS:
Drug: Verapamil — Patients in groupe A require verapamil initiation as a preventive treatment and patients in group B are patients already undergoing a verapamil treatment for their Cluster Headache.
  The doses of verapamil are increased for the patients in group A, after a clinical examination an electrocardiogram, and a blood test.

SUMMARY:
Verapamil is a calcium channel blocker widely used to treat cardiovascular diseases however it is also the first line treatment in the prevention of cluster headaches. In France, its prescription in that indication is based on compliance with the Temporary Recommendation for Use (RTU) that insists on the possible the cardiac side effects that can occur as the doses required for cluster headache are significantly higher than the doses used in cardiology.

ELIGIBILITY:
Inclusion Criteria:

* patient 18 years old, and older
* patient suffering from Cluster Headache (according to the l'ICHD-3 diagnostic criterias)
* patients affiliated to the social security
* patient that has given his full written consent to participate in the study
* female patients participating in the study must be using an efficient contraception for more than 1 month prior to the beginning of the study

Exclusion Criteria:

* patient presenting contraindications to the use of verapamil
* patient observing a treatment with ivabradine (Procoralan®), bétablockers, colchicine, l'esmolol, triazolam, quinidine.
* patient under justicial protection
* patient breastfeeding, or pregnant
* patient suffering from a neuromuscular transmisson disease
* patient with a pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2027-09-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the atrioventricular block when verapamil is used in prevention of Cluster Headache. | 27 months
  Occurrence of the ratio of patients presenting a first degree atrioventricular block

SECONDARY OUTCOMES:
Description of the different atrioventricular conduction abnormities and their incidence | 27 months
  Study of ECG results
Evaluation of the plasmatic concentration of verapamil and its metabolite (nor verapamil) in parallel with the occurrence of conduction abnormalities detected by electrocardiogram | 27 months
  Plasmatic concentration of verapamil and its metabolite (nor verapamil) dosed at each visit
Relation between pharmacokinetic/ pharmacodynamics of verapamil and the appearance of conduction abnormalities to determinate the maximal tolerated dose of verapamil. | 27 months
  The maximal tolerated dose of verapamil will be determined thanks to correlation between ECG results and Pharmacocinetics and pharmacodynamics

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Nice, Nice, CHUN
  - AP-HP Hôpital la Timone, Marseille

IPD SHARING:
Plan to Share IPD: No
No data sharing plan ahs been established